CLINICAL TRIAL: NCT03227965
Title: Immunosuppression's Long Term Impact on Anti-tumoral Oversight in Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ELITE
Record Dates: First submitted 2017-06-23; First posted 2017-07-24 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Kidney Transplant; Complications
Keywords: cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ELITE (Other)
  Interventions: Biological: Immune cells population assesment

INTERVENTIONS:
Biological: Immune cells population assesment — T lymphocytes population description through blood, urine and faeces samples

SUMMARY:
Cancer is a well known complication about long term transplantation. Cancer outcomes are due to the immunosuppressive treatment that prevents transplanted people from rejection. By lowering the effectiveness of the immune system, immune cells are no longer able to seek and destroy cancer cells.

The goal here is to study immunes cells population of people that were transplanted 10 years ago and are now treated either by a corticosteroid - azathioprine association, or only by cyclosporine A.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* Patients with kidney transplantation for 10 year
* Patients with stable renal function (less than 20% creatinine variation during the last 12 months)
* Patients treated either by a corticosteroid - azathioprine association or cyclosporine A
* Patients giving his agreement
* Patients legally free

Exclusion Criteria:

* Patients under 18
* Patients under legal protection
* Pregnant women, or of age to get pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Immune cells study | 12 months
  Study 2 types of T lymphocytes (by flow cytometry) that are suspected to be responsible of the graft non rejection and the cancer outcome, treated by corticosteroid - azathioprine association or cyclosporine A

SECONDARY OUTCOMES:
bacteria study | 12 months
  Study the modification of the intestinal bacteria population that might led to an "operational tolerance", depending on the immunosuppressive treatment : the DNA will be extracted from the faeces and a typing will be carried out by Polymerase Chain Reaction
cancer incidence | 12 months
  Assess cancer incidence, on a population of people with kidney transplantation (since 10 years) : observation of adverse events during visits

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Poitiers, Poitiers, France